CLINICAL TRIAL: NCT01977820
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized, 2-Arm Phase IIa Pilot Trial Assessing the Effect of Sapropterin on Cognitive Abilities in Young Adults With Phenylketonuria
Brief Title: Sapropterin on Cognitive Abilities in Young Adults With Phenylketonuria
Acronym: SIGNAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR 700773-004; 2010-024311-13 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; Sapropterin; Placebo; Cognitive Abilities; Kuvan®
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sapropterin (Experimental)
  Interventions: Drug: Sapropterin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sapropterin — Sapropterin tablets will be administered orally once daily at a dose of 20 milligram per kilogram (mg/kg) during both the 2-Week response test period and 24-Week study period.
  Other Names: Kuvan®
  Arms: Sapropterin
Drug: Placebo — Sapropterin tablets will be administered orally once daily at a dose of 20 milligram per kilogram (mg/kg) during both the 2-Week response test period and Placebo tablets matching to sapropterin will be administered orally once daily during the 24-Week study period.
  Arms: Placebo

SUMMARY:
This is a Phase 2a multicenter, double-blind, placebo-controlled, randomized, 2-arm pilot trial designed to assess the effect of sapropterin on cognitive abilities in young adults with Phenylketonuria (PKU) over a 26-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given before any trial-related activities are carried out
* Women or men with documented PKU diagnosed by at least two phenylalanine levels equal or greater than 600 micromole per liter (mcmol/L)
* For women of childbearing potential: a negative urine pregnancy test is required at screening and willingness to use a highly effective method of contraception is required during the study and follow-up periods
* Aged greater than or equal to (>=) 18 to 29 years, inclusive
* Mean blood phenylalanine levels 600 to 1000 mcmol/L during 12 months preceding inclusion in the study. The mean should be calculated from at least 3 blood phenylalanine values over the last 12 months. Screening blood phenylalanine level can be one of these values. There should be at least one value dated between Month -12 and -6 before Screening and at least one value dated between Month -6 and Screening
* An intelligence quotient (IQ) score greater than or equal to 85, assessed a maximum of 2 years before screening with an age-appropriate Wechsler scale. If no IQ test result is available, IQ testing must be performed as part of Screening using an age-appropriate Wechsler scale before the subject can be included
* Subjects willing to comply with all study procedures, including willingness to continue current dietary recommendations during the whole trial duration

Exclusion Criteria:

* Subjects with tetrahydrobiopterin (BH4) deficiency
* Previous exposure to sapropterin or BH4 for greater than 30 days (or exposure to sapropterin or BH4 for less than or equal to 30 days but within the previous 6 months prior to Screening visit)
* Subjects who, according to the Investigator, will not be able to comply with study procedures and computerized neuropsychological testing
* Any significant illness which, according to the Investigator, might preclude participation in the study (including neurological disease, cardio-vascular disease, history of seizure, predisposition to convulsions, renal or hepatic insufficiency, and active malignancy)
* Any significant illness, medication or substance abuse which, according to the Investigator, might affect cognitive function and cognitive testing (for example, significant visual or motor impairment, history of major head trauma, history of stroke, alcoholism, drug dependency, psychological disorder requiring chronic use of psychotropic medications such as anxiolytics, antidepressants, antipsychotic medication, mood stabilizers, and hypnotics)
* Concomitant forbidden medication as described in the Kuvan® Summary of Product Characteristics, namely, inhibitors of dihydrofolate reductase (for example, methotrexate, trimethoprim), medications that are known to affect nitric oxide synthesis (for example, glyceryl trinitrate, isosorbide dinitrate, sodium nitroprusside, molsidomin, phosphodiesterase type 5 inhibitors, and minoxidil), and levodopa, as it may cause increased excitability and irritability
* Known hypersensitivity to sapropterin or any ingredients in the product's formulation, or to other approved or non-approved formulations of BH4
* Subjects who have undergone cognitive neuropsychological testing similar to that to be performed as part of this trial with the following time limits: tasks with limited practice effect performed in the last 6 months, and tasks with important practice effect (such as tasks involving development of strategies) performed in the year preceding inclusion in the trial. Whether a task falls into one or the other category is left to Investigator judgment
* Female subjects who are pregnant or in the lactation period
* Subjects currently participating to another clinical trial or who participated in a previous clinical trial within 30 days prior to screening
* Legal incapacity or limited legal capacity

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — BioMarin Pharmaceutical
Locations (2):
- Research Site, Bologna, Italy
- Research site, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): 24 Feb 2014/12 Aug 2014. Study premature termination date: 07 Nov 2014; Subjects were randomized at 2 study centers.
Pre-assignment Details: A total of 10 subjects were screened and 7 subjects were included in the 2-Week response test period. Out of 7 subjects, only 2 subjects were responders and they were enrolled and randomized to receive study drug into the 24-Week study period.
Groups:
- Sapropterin: Subject was administered with 20 milligram per kilogram (mg/kg) sapropterin tablets orally once daily during the 2-week response test period. The subject upon completing the 2-Week response test period was randomized to receive sapropterin during the 24-week study period. The subject underwent the study assessments and procedures according to the study protocol until the study was terminated by the Sponsor.
- Placebo: Subject was administered with 20 mg/kg sapropterin tablets orally once daily during the 2-week response test period. The subject upon completing the 2-Week response test period was randomized to receive placebo tablets matching to sapropterin orally once daily during the 24-week study period. The subject underwent the study assessments and procedures according to the study protocol until the study was terminated by the Sponsor.
Period: Overall Study
Arm/Group | Sapropterin | Placebo
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Sponsor terminated the study | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the subjects randomized into 24-Week study period and received least 1 dose of study drug.
Groups:
- Sapropterin: Subject was administered with 20 mg/kg sapropterin tablets orally once daily during the 2-week response test period. The subject upon completing the 2-Week response test period was randomized to receive sapropterin during the 24-week study period. The subject underwent the study assessments and procedures according to the study protocol until the study was terminated by the Sponsor.
- Total: Total of all reporting groups
Arm/Group | Sapropterin | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Number; unit: Subjects]
  >=18 to 29 Years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs), Serious AEs (SAEs), AEs Leading to Death and AEs Leading to Discontinuation
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Screening up to 24 weeks + 4-week follow-up
Population: The safety analysis population included all the randomized subjects who received at least one dose of study treatment.
Measure: Number; unit: Subjects
Groups:
- Sapropterin: Subject was administered with 20 mg/kg sapropterin tablets orally once daily during the 2-week response test period. The subject upon completing the 2-Week response test period was randomized to receive sapropterin during the 24-week study period. The subject completed the study according to the study protocol until the study was terminated by the Sponsor.
- Placebo: Subject was administered with 20 mg/kg sapropterin tablets orally once daily during the 2-week response test period. The subject upon completing the 2-Week response test period was randomized to receive placebo tablets matching to sapropterin orally once daily during the 24-week study period. The subject completed the study according to the study protocol until the study was terminated by the Sponsor.
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 1 | 1
Subjects
  AEs | 1 | 0
  SAEs | 0 | 0
  AEs leading to death | 0 | 0
  AEs leading to discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening up to 24 weeks + 4-week follow-up
Arm/Group | Sapropterin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin (N=1) | Placebo (N=1)
Headache (Nervous system disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued by the Sponsor due to severe enrolment difficulties as a consequence of the limited availability of treatment naïve patients with a diagnosis of phenyl ketonuria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All written or oral publications and/or information related to Study and/or results of Study should be submitted at first in writing to Sponsor at least 30 working days for publication and 15 working days for brief review, abstract before planned date of submission. If Sponsor is filing a patent application on Study results, Sponsor can delay its authorization for publication/communication of Study results to Investigator and/or Research Centre until date of international registration of patent.